CLINICAL TRIAL: NCT03976817
Title: Supra-annular Aortic Valve Replacement: Surgical Techniques and Early Outcomes
Brief Title: Aortic Valve Replacement Above the Aortic Annulus (SA-AVR) With the Carpentier-Edwards Magna-Ease Bioprosthesis
Acronym: SA-AVR
Status: Completed | Type: Observational
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Other Study IDs: TPS 59185
Record Dates: First submitted 2019-05-28; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-05

CONDITIONS: Aortic Valve Disease; Prosthesis; Cardiac, Heart, Functional Disturbance as Result
Keywords: bioprosthesis; surgery; supra-annular
MeSH Terms: conditions — Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SA-AVR group: Patients who underwent the supra-annular aortic valve replacement (SA-AVR) technique in our institution between December 2010 and December 2017 were retrospectively reviewed.
  Interventions: Procedure: aortic valve replacement

INTERVENTIONS:
Procedure: aortic valve replacement — After median sternotomy, cardiopulmonary bypass (CPB) was established between the ascending aorta and the right atrium. The aorta was cross-clamped and a high potassium warm cardioplegia was infused and repeated every 15 minutes. The aortotomy was made above the sinuses and the aortic valve was removed. The prosthesis was chosen one size larger than the maximal sizer that could be inserted, which was also used to determine the appropriate height for insertion of the sutures along the wall of the non-coronary sinus.

SUMMARY:
Surgical valve replacement is commonly performed in patients with severe aortic valve disease. In small aortic annulus, implantation of bioprosthetic valves can be associated with limited functional capacity. To avoid this condition, we changed our surgical technique to implant a larger bioprosthesis. Briefly, the prosthesis is sutured to the aortic annulus along the left and right coronary sinuses, and in a supraannular position along the noncoronary sinus, therefore allowing us to insert a prosthetic valve with a one-size larger diameter than the native aortic annulus.

DETAILED DESCRIPTION:
Surgical aortic valve replacement (AVR) is recommended for severe aortic valve disease. Bioprosthesis remains the substitute of choice for elderly patients. However, it may be associated with patient-prosthesis mismatch particularly for patients with small aortic annulus. Moreover, "valve-in-valve" transcatheter aortic valve replacement (TAVR) has become a suitable therapeutic option for bioprosthesis structural degeneration, especially in patients with high surgical risk. It is therefore of great importance to implant the widest bioprosthesis as possible at the first AVR. The investigators report a surgical technique allowing the implantation of a larger bioprosthesis in patients with small aortic annulus: the supra-annular aortic valve replacement (SA-AVR) above the aortic annulus. The investigators analyzed the postoperative outcomes of the SA-AVR technique using the Perimount Magna Ease (Carpentier-Edwards, Irvine, California) bioprosthesis.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years who underwent a suprannular implantation of the Carpentier Edwards Magna Ease bioprosthetic valve between January 2010 and December 2017 in our institution, whatever the aetiology of the aortic valve disease.

Exclusion Criteria:

* patients younger than 18 years, patients who received a different bioprosthesis valve in the aortic position, patients who were lost of follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent aortic valve replacement in our institution
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | Hospital discharge, an average 10 days

SECONDARY OUTCOMES:
Functional status | 1 year after the surgery
  New York Heart Association functional class (from I to IV)

CONTACTS AND LOCATIONS:
Overall Officials: Elie Fadel, MD PhD, Study Chair — Marie Lannelongue Hospital
Locations (1):
- Hopital Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No